CLINICAL TRIAL: NCT02887092
Title: Determinants of Functional Ability and Perceived Health, and Interaction With Multimorbidity in Hip and Knee Osteoarthritis
Brief Title: Determinants of Functional Ability, Perceived Health, and Interaction With Multimorbidity in Hip and Knee Osteoarthritis
Acronym: PRO-ART
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: University of Lorraine (Other); University of Paris 5 - Rene Descartes (Other)
Responsible Party: Principal Investigator, GUILLEMIN Francis, MD, professor, Central Hospital, Nancy, France
Other Study IDs: PRO-ART
Record Dates: First submitted 2016-08-25; First posted 2016-09-01 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Osteoarthritis
Keywords: health determinants; epidemiology; maintaining autonomy; psychology; osteoarthritis; perceived health
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Hip and knee osteoarthritis (OA) is an important health problem with a high prevalence and significant consequences on functional ability, perceived health, restriction of autonomy and handicap. The weight of multimorbidities and their interaction on functional ability and perceived health are left unexplored. This project will rely on the cohort KHOALA, representative, multiregional, of 881 prevalent cases (symptomatic hip and knee OA).

Main objective:

* to describe the evolution over time of pain, functional ability, social participation and quality of life in subjects with hip and knee OA
* to identify prognosis factors of disease evolution (socio-demographic, clinical, and other health parameters)
* to determine interactions with comorbidities, other personal and environmental factors (ICF model).

Concurrent objective: to improve measurement of perceived health specific to hip and knee OA by the OAKHQOL by improving its metrologic performances based on item response theory.

Task 1: To prepare an improved measurement scale, available as a judgment criteria for the 3rd year of cohort follow up, over the april 2010-march 2012 period, the mini-OAKHQOL Task 2: Evaluation of the cohort in 2010-2012 (year 3 of follow up) in a repeated measure design to best assess the evolution of perceived health and functional ability over time, and to identify stability of deterioration of autonomy. Perspectives: This project targets to provide public health deciders with information of good quality to help them manage determinants of perceived health in OA subjects, as essential factors to health care resource utilization in their various modalities.

ELIGIBILITY:
Inclusion Criteria:

* hip or knee osteoarthritis (tibiofemoral), uni or bilateral, symptomatic, with confirmed diagnosis according to American College of Rheumatology ACR and European League Against Rheumatism (EULAR)
* Kellgren and Laurence radiological stage at least 2

Exclusion Criteria:

* knee or hip prosthesis on painful joint
* preceding osteotomy
* serious comorbidity (affecting quality of life, or leading to a high care consumption)
* according to X-ray : knee pain with isolated patello-femoral osteoarthritis (i.e without an associated tibiofemoral osteoarthritis)
* other pathology on knee or hip
* adults getting a legal protection or with the incapacity to give their consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with hip or knee osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 881 (Actual)
Dates: Start 2007-04; Primary Completion 2009-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
change in quality of life | 3 years

SECONDARY OUTCOMES:
comorbidity | 3 years
  Functional comorbidity index
change in functional ability | 3 years
  Womac score
change in pain | 3 years
  VAS

CONTACTS AND LOCATIONS:
Overall Officials: Francis Guillemin, MD, PhD, Principal Investigator — CHRU Nancy

IPD SHARING:
Plan to Share IPD: Yes